CLINICAL TRIAL: NCT01881633
Title: A Dose Block-randomized, Double-blind, Placebo-controlled, Single Dosing, Dose-escalation Phase I Clinical Trial to Evaluate the Tolerability, Safety, and Pharmacokinetics of ISU302 in Healthy Volunteers
Brief Title: A Study of the Tolerability, Safety, and Pharmacokinetics of ISU302 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ISU Abxis Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: ISU-002
Record Dates: First submitted 2013-06-14; First posted 2013-06-19 (Estimated); Last update posted 2013-06-19 (Estimated); Status verified 2013-06

CONDITIONS: Gaucher Disease
Keywords: gaucher disease, imiglucerase, ISU302
MeSH Terms: conditions — Gaucher Disease

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (4):
- ISU302 (Experimental): 15 U/kg I.V. injection
  Interventions: Drug: ISU302
- ISU302 30 U/kg (Experimental): Drug ISU302 I.V. injection
  Interventions: Drug: ISU302
- ISU302 60 U/kg (Experimental): Drug ISU302 I.V. injection
  Interventions: Drug: ISU302
- Placebo (Placebo Comparator): ISU302 Placebo I.V. injection
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ISU302
  Arms: ISU302; ISU302 30 U/kg; ISU302 60 U/kg
Drug: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess the safety, tolerability, and pharmacokinetics of single dosing study with three ascending dose cohorts of ISU302 in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male volunteers, aged between ≥ 20 and ≤ 45 years old
* Weight ≥ 50, with calculated body mass index of 17 and 25 kg/m2

  * BMI = (Weight [kg])/(height [m])2
* Subject is informed of the investigational nature of this study and voluntarily agrees to participate in this study and comply with the relevant instructions in written
* Considered ineligible through screening test (such as medical history, physical examination, ECG, safety laboratory test) performed within 35 days prior to study start (dosing of investigational products)

Exclusion Criteria:

* With symptoms indicating acute diseases within 28 days prior to start of study (dosing of investigational product)
* History or presence of clinically significant and active cardiovascular, respiratory, renal, endocrine, hematological, gastrointestinal, central nervous system, psychiatric disorder, autoimmune disease, or malignant tumor
* Any medical history that may affect drug absorption, distribution, metabolism and excretion(e.g., inflammatory gastric disease, gastric or intestinal ulcer, hepatic or renal disease)
* With presence of clinically significant allergic disease (including mild allergic rhinitis or allergic dermatitis which does not need medication)
* With presence of clinically significant hypersensitivity to any drugs
* With hemolytic anemia, anemia due to blood loss (Hb < 14g/dL and Hct <42%)
* With the results of safety laboratory test

  1. AST (Aspartate Transaminase) or ALT (Alanine Transaminase) > 1.5 times of upper normal limit
  2. Total bilirubin > 1.5 times of upper normal limit
* Subject who has immune deficiency or medication with immune suppressants
* Participation in other clinical study within 60 days prior to start of study (dosing of investigational products)
* Use of any drugs, possibly affecting drug metabolizing enzymes, within 1 month prior dosing, or any drugs, possibly affecting the results of clinical trial within 10 days or use of drug was not passes 5 x half-life of drug
* Donated whole blood within 60 days, or transfused within 20 days before the study
* History of alcohol abuse (> 14 units/week) and the subject could not stop drinking alcohol beverage during study period
* Heavy smoker (>10 cigarettes/day) or the subject could not stop smoking during study period
* Unwillingness or inability to follow the procedures outlined in the protocol
* Positive in pregnancy test in urine and unwilling to follow contraception during study period and following 3 months (for female subjects).

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2010-10; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability | From Screening to Day 5 post-dose
  Evaluation for safety data by treatment group/ Confirmative evaluation for serious adverse drug reaction/ Descriptive statistics (arithmetic mean and standard deviation) for quantitative analysis and evaluation of change from baseline/ Frequency counts for qualitative categorization of safety data
  Parameters:
  * Adverse events including subjective/objective symptoms
  * Physical examination
  * 12-lead ECG
  * Vital signs
  * Local tolerability test
  * Clinical laboratory test: Hematology, Coagulation, Blood Chemistry, Urinalysis
  * Immunogenicity

SECONDARY OUTCOMES:
Pharmacokinetics | Day1
  Pharmacokinetic Parameter assessment using non-compartmental analysis from the concentration-time data/ Summary of Pharmacokinetic parameters by treatment group using descriptive statistics/ Dose proportionality
  Parameters: Cmax, AUCt, AUCinf, Tmax, t1/2, Clearance, Vd, MRTr